CLINICAL TRIAL: NCT03386669
Title: Novel Neuroimage Study in Tauopathies With Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201601674A0
Record Dates: First submitted 2017-08-14; First posted 2017-12-29 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Parkinsonism
Keywords: 18F-THK5351 PET; Tauopathies
MeSH Terms: conditions — Parkinsonian Disorders; Tauopathies | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-18 AV-45 THK-5351 (Experimental): F-18 AV-45 THK-5351 imaging
  Interventions: Drug: F-18

INTERVENTIONS:
Drug: F-18 — Totally 60 subjects age 20-80 including 20 subjects with a diagnosis of PD,PSP,and CBS. For disease subjects, caregiver should be able to report activities of daily living and their mental status. Patient should be able to give informed consent or have a caregiver give consent with subject assent.
  Other Names: F-18 THK-5351; F-18 AV-45

SUMMARY:
The aims of this study are: 18F-THK5351 PET(Positron Emission Tomography) can defect the tau burden in PSP(Progressive Supranuclear Palsy) and CBS (Corticobasal syndrome)correlating with the known NFT(neurofibrillary tangles) topology of those diseases, 18F-THK5351 PET will differentiate subjects with suspected tauopathy due to PSP and CBS from subjects with suspected synucleinopathy due to idiopathic PD(Parkinson's disease). The distribution of PHF(paired helical filament) tau burden will correlate with specific motor and cognitive features of PSP and CBS; and regional PHF tau burden will be associated with cortical thinning. Together, these efforts will establish the potential for developing 18F-THK5351 PET imaging as a biomarker and diagnostic tool for the parkinsonian tauopathies.

ELIGIBILITY:
Inclusion Criteria:

1. 20 subjects with a diagnosis of PD whom must:

   * Age ranges from 20-80 years
   * Patients should be fulfilled "UK(United Kingdom ) Parkinson's Disease Society Brain Bank Criteria for the diagnosis of PD", 2.11.1 Appendix I, (27)
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
2. 20 subjects with a diagnosis of PSP whom must:

   * Age ranges from 20-80 years
   * Patients fulfill the criteria of NINDS-SPSP(National Institute of Neurological Disorders and Stroke / Society for PSP) clinical criteria for the diagnosis of PSP "as possible" or "probably" PSP, 2.11.2 Appendix II, (28)
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
3. 20 subjects with a diagnosis of CBS whom must:

   * Age ranges from 20-80 years
   * Patients should be fulfilled the "Mayo Clinic proposed criteria for the diagnosis for corticobasal syndrome" , 2.11.3 Appendix III, (29)
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

Exclusion Criteria:

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases
3. Major psychiatric disorders, drug or alcohol abuse and major depression
4. Pregnant women or breast- feeding women
5. Patients in whom MRI was contraindicated
6. History of severe allergic or anaphylactic reactions particularly to the tested drugs
7. Indication of impaired liver function as shown by an abnormal liver function profile at screening (eg. repeated values of aspartate aminotransferase [AST(aspartate aminotransferase)] and alanine aminotransferase [ALT(Alanine aminotransferase)] ≧ 3X(3 Times) the upper limit of normal values)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
To establish Tau image pattern for Tauopathies with parkinsonism. | YEAR ONE
  Use ANOVA analysis(Analysis of variance) to significant differences in regional 18F-THK-5351 uptake between PSP, CBS and PD groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan, Guishan Dist, Taiwan